CLINICAL TRIAL: NCT00056823
Title: A Phase I/II, Single-Masked, Multicenter Study of the Safety, Tolerability, and Efficacy of Multiple-Dose Intravitreal Injections of rhuFab V2 in Combination With Verteporfin (Visudyne(R)) Photodynamic Therapy in Subjects With Neovascular Age Related Macular Degeneration
Brief Title: Intravitreal Injections of rhuFab V2 in Combination With Visudyne in Subjects With Age Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FVF2428g
Record Dates: First submitted 2003-03-24; First posted 2003-03-26 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Age-Related Maculopathy
Keywords: AMD
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

INTERVENTIONS:
Drug: rhuFab V2 (ranibizumab)

SUMMARY:
The primary purpose of this study is to determine if injections of rhuFab V2 into the eye in combination with verteporfin photodynamic therapy (PDT) is a safe and efficacious treatment for patients with age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age >=50 years
* Eligibility for treatment with PDT using verteporfin in the study eye according to the Visudyne(R) product labeling
* Treatment with verteporfin anticipated or expected
* Primary or recurrent subfoveal choroidal neovascularization (CNV) lesions secondary to AMD in the study eye
* A classic CNV component (well-demarcated hyperfluorescence boundaries in the early phase of the fluorescein angiogram) that is >=50% of the total lesion area
* Total lesion size >=5400 um in greatest linear dimension (GLD)
* Best corrected visual acuity, using ETDRS charts, of 20/40 to 20/320 (Snellen equivalent) in the study eye

Exclusion Criteria:

* Treatment with verteporfin in the study eye less than 3 months preceding Day 0
* Treatment with verteporfin in the non-study eye less than 7 days preceding Day 0
* More than three prior treatments with verteporfin PDT in the study eye within 12 months preceding Day 0
* Prior treatment with external-beam radiation therapy or transpupillary thermotherapy in the study eye
* Previous participation in a clinical trial (for either eye) involving antiangiogenic drugs (pegaptanib, rhuFab V2, anecortave acetate, protein kinase C inhibitors, etc.) Previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection or device implantation) in the study eye
* Previous subfoveal focal laser photocoagulation in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1 month preceding Day 0
* History of vitrectomy, submacular surgery, or other surgical intervention for AMD in the study eye
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals studies)
* Subretinal hemorrhage in the study eye that involves the center of the fovea, if the size of the hemorrhage is either >=50% of the total lesion area or >=1 disc area in size
* Subfoveal fibrosis or atrophy in the study eye
* Clinical or angiographic evidence of retinal angiomatous proliferation in the study eye, if there is also no angiographic evidence of classic CNV
* CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia
* Retinal pigment epithelium tear involving the macula in the study eye
* Any concurrent intraocular condition (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, either could require medical or surgical intervention during the 24-month study period to prevent or treat visual loss that might result from that condition, or if allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of best corrected visual acuity over the 24-month study period
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye. Infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia or absence of the posterior capsule in the study eye
* Spherical equivalent of the refractive error in the study eye demonstrating more than -8 diopters of myopia
* Intraocular surgery (including cataract surgery) on the study eye within 1 month preceding Day 0
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure >=30 mmHg despite treatment with anti-glaucoma medication)
* Premenopausal women not using adequate contraception
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications.
* Current treatment for active systemic infection
* Contraindications to verteporfin photodynamic therapy (as determined by the investigator)
* History of allergy to fluorescein, not amenable to treatment
* Inability to dilate pupils to >=6 mm in diameter
* Inability to comply with study or follow up procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168
Dates: Start 2003-03; Study Completion 2005-12 (Actual)

REFERENCES:
- [Derived] Xu L, Lu T, Tuomi L, Jumbe N, Lu J, Eppler S, Kuebler P, Damico-Beyer LA, Joshi A. Pharmacokinetics of ranibizumab in patients with neovascular age-related macular degeneration: a population approach. Invest Ophthalmol Vis Sci. 2013 Mar 5;54(3):1616-24. doi: 10.1167/iovs.12-10260. PMID 23361508
- [Derived] Antoszyk AN, Tuomi L, Chung CY, Singh A; FOCUS Study Group. Ranibizumab combined with verteporfin photodynamic therapy in neovascular age-related macular degeneration (FOCUS): year 2 results. Am J Ophthalmol. 2008 May;145(5):862-74. doi: 10.1016/j.ajo.2007.12.029. Epub 2008 Mar 5. PMID 18321465